CLINICAL TRIAL: NCT02338492
Title: A Prospective, Multi-Center Study of the IlluminOss® Photodynamic Bone Stabilization System for the Treatment of Impending and Actual Pathological Fractures in the Humerus From Metastatic Bone Disease
Brief Title: Safety and Efficacy Study of Treatment of Pathological Fractures in Humerus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IlluminOss Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-03-PATHOLHUM-02
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Humerus Fracture Metastatic Bone Disease

ARMS (1):
- Photodynamic Bone Stabilization System (Experimental): Photodynamic Bone Stabilization System (PBSS) is comprised of an inflatable, thin walled polyethylene terephthalate (PET; Dacron™) balloon mounted on an insertion catheter. This balloon catheter system is designed to deliver the monomer cement to the fracture site via the medullary canal of the bone
  Interventions: Device: Photodynamic Bone Stabilization System

INTERVENTIONS:
Device: Photodynamic Bone Stabilization System — Treatment of impending and actual pathological fractures of the humerus

SUMMARY:
This study will collect safety and performance data of the Photodynamic Bone Stabilization System (PBSS) when used for the treatment of fractures of the humerus secondary to metastatic cancer.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open label study to evaluate the Photodynamic Bone Stabilization System (PBSS) when used for the treatment of painful impending and actual fractures of the humerus secondary to metastatic malignancy.

ELIGIBILITY:
Inclusion Criteria:

- General Inclusion Criteria

1. Skeletally mature adult males and females 18 years of age or older.
2. Impending or actual pathological fracture of the humerus, secondary to metastatic bone disease.
3. Females: neither pregnant nor intending to become pregnant during the course of the study, defined as:

   1. Postmenopausal for at least 1 year OR
   2. Documented oophorectomy or hysterectomy
   3. Surgically sterile OR
   4. If of childbearing potential, must be practicing double-barrier method of birth control, be willing to avoid pregnancy for the period of study participation and have a negative pregnancy test at screening
4. Patient, or his/her legally authorized representative, is able to understand and provide informed consent.
5. Willing and able to comply with post-operative treatment protocol and follow-up visit schedule.
6. VAS Pain Score > 60mm on 100mm scale.

   -Impending Fracture-Specific Inclusion Criteria
7. Documented presence of at least one metastatic lesion of the humerus.
8. Mirels Criteria Score ≥ 8. (specific to the target humeral lesion and subject to minimum VAS score requirements)
9. Destruction of cortical bone at impending fracture site > 50%.

   -Actual Fracture-Specific Inclusion Criteria
10. Fracture is closed, Gustilo Type I or II.

Exclusion Criteria:

- General Exclusion Criteria

1. Primary tumor (osteogenic origin, etc.) at site.
2. Impending or actual fracture at any other location that, in the Investigator's opinion, would preclude ability to assess pain and/or function in the target humerus.
3. Active or incompletely treated infections that could involve the device implant site.
4. Distant foci of infection that may spread to the implant site.
5. Allergy to implant materials or dental glue.
6. In the investigator's judgment, functional deficit in the target humerus with an etiology other than bone metastases (e.g. due to vascular insufficiency).
7. In the investigator's judgment, focal neurologic deficit as a result of metastases in the brain, spine, or other central nervous system disorders.
8. Uncooperative patients, or patients who are incapable of following directions (for example, as a consequence of a neurological or psychiatric disorder).
9. Prisoner

   -Impending Fracture-Specific Exclusion Criteria
10. Mirels Score < 8 (specific to target humeral lesion).
11. Destruction of cortical bone at impending fracture site < 50%.
12. Prior surgery and/or prior fracture of affected site.
13. Any articular component to impending fracture site.

    -Actual Fracture-Specific Exclusion Criteria
14. Open fractures with severe contamination.
15. Extremely comminuted fractures where insufficient holding power of the balloon on the intramedullary canal is probable.
16. Patients whose intramedullary canal at site of fracture measures smaller than the diameter of the sheath provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Stanford School of Medicine, Redwood City, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Physicians, Pittsburgh, Pennsylvania
  - University Orthopedics Inc., Providence, Rhode Island
  - Marshall University, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Photodynamic Bone Stabilization System (PBSS): The PBSS is comprised of an inflatable, thin walled polyethylene terephthalate (PET; Dacron™) balloon mounted on an insertion catheter. This balloon catheter system is designed to deliver the monomer cement to the fracture site via the medullary canal of the bone
  IlluminOss® Photodynamic Bone Stabilization System (PBSS): Treatment of impending and actual pathological fractures of the humerus
Period: Overall Study
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Started | 81
Enrolled | 81
Device Implanted | 79
Treatment Failure | 2
Completed | 36
Not Completed | 45
Not completed — Death | 32
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 4
Not completed — Reason not captured above | 6

BASELINE CHARACTERISTICS:
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 68
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81
Actual Bone Fracture Characteristics - Location of Target Fracture [Count of Participants; unit: Participants] — Population: Subjects with Actual Bone Fracture
  Participants
    number analyzed (Participants) | 49
    Left Humerus | 24
    Right Humerus | 25
Actual Bone Fracture Characteristics - Location [Count of Participants; unit: Participants] — Population: Subjects with Actual Bone Fracture
  Participants
    number analyzed (Participants) | 49
    Proximal | 25
    Diaphyseal | 20
    Distal | 4
Actual Bone Fracture Characteristics - AO Classification [Count of Participants; unit: Participants] — Classification system of fractures. 11 is the proximal humerus, 12 is the humeral shaft, and 13 is the distal humerus. For the proximal humerus, A is an extra-articular unifocal fracture, B is an extra-articular bifocal fracture and C is an articular fracture. For the humeral shaft, A is a simple fracture, B is a wedge fracture and C is a complex fracture. For the distal humerus, A is an extra articular fracture, B is partial articular fracture and C is a complete articular fracture. These are further classified as 1, 2, 3 with the higher number indicating a more complex fracture. Population: Subjects with Actual Bone Fracture
  Participants
    number analyzed (Participants) | 49
    11-A1 | 1
    11-A2 | 6
    11-A3 | 5
    12-A1 | 7
    12-A2 | 12
    12-A3 | 5
    12-B1 | 3
    12-B2 | 7
    12-C3 | 1
    NA | 1
    Unknown | 1
Actual Bone Fracture Characteristics - Gustilo Grading of Soft Tissue [Count of Participants; unit: Participants] — Soft tissue grading. It ranges from Type I (wound < 1 cm) to Type III C (vascular injury requiring vascular repair), with the wound damage getting more severe as the type increases. A closed fracture does not have any soft tissue damage. The grading system considers the energy of the injury, the wound size, amount of soft tissue damage, contamination, fracture pattern, periosteal stripping, skin coverage, neovascular injury and antibiotic use. Population: Subjects with Actual Bone Fracture
  Participants
    number analyzed (Participants) | 49
    Closed Fracture | 46
    Type I | 3
Impending Bone Fracture Characteristics - Location of Target Fracture [Count of Participants; unit: Participants] — Population: Subjects with Impending Bone Fracture
  Participants
    number analyzed (Participants) | 32
    Left Humerus | 14
    Right Humerus | 18
Impending Bone Fracture Characteristics - Location [Count of Participants; unit: Participants] — Population: Subjects with Impending Bone Fracture
  Participants
    number analyzed (Participants) | 32
    Proximal | 22
    Diaphyseal | 9
    Distal | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Change in VAS score from baseline. VAS is measured on a scale range from 0-100mm with 0 (no pain) to 100 (worst imaginable pain).
Time Frame: Baseline and 90 days
Population: Number of subjects who had a Day 90 visit
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 56
units on a scale | -52.7 (3.62)
Statistical Analysis 1: Comparison: Photodynamic Bone Stabilization System (PBSS); Null hypothesis: Mean improvement in VAS over 90 days <= 53.8 (i.e. 80% of reference based on historical control data). The study was powered to 80% with 68 evaluable subjects, a standard deviation of 13.3 at each visit, a true mean improvement from baseline VAS across post-baseline visits of 57 and a within-patient correlation of VAS of 0.4. The historical control data comes from 4 selected articles (Gregory et al. 2011, Kim et al. 2011, Deschamps et al. 2012, and Pretell et al. 2010); Test type: Superiority; p = 0.615, Mixed Models Analysis — P-value not adjusted for multiple comparisons as the second co-primary endpoint will only be tested if the p-value for VAS improvement is <0.05; Mixed model repeated measures (MMRM) model employed, including the baseline VAS score. Missing values will be imputed

2. Primary Outcome: Change in Function
Description: Change in Revised Musculoskeletal Tumor Society Rating Scale for Upper Extremity (MSTS). MSTS score is a six-item scale. It ranges from 0 to 30. Higher score is associated with better function. Scores were divided by 30 and multiplied by 100 to facilitate interpretation.
Time Frame: Baseline and 90 days
Population: Subjects who had 90 Day data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 52
units on a scale | 39.23 (2.929)

3. Primary Outcome: Summary of Clinical Safety Success
Description: No serious device related complications, no additional surgical interventions, and no device fracture, migrations, mal-alignment or loss of reduction or fixation
Time Frame: Up to Day 7-14, Up to Day 30, Up to Day 90, Up to Day 180, Up to Day 360
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Participants
  Up to D7-14 : No serious dev rel complications | 81
  Up to D7-14 : No additional surgical intervention | 81
  Up to D7-14 : No device fracture, migration | 80
  Up to D7-14 : Safety Success | 80
  Up to D30 : No serious dev rel complications | 80
  Up to D30 : No additional surgical intervention | 80
  Up to D30 : No device fracture, migration | 78
  Up to D30 : Safety Success | 78
  Up to D90 : No serious dev rel complications | 78
  Up to D90 : No additional surgical intervention | 80
  Up to D90 : No device fracture, migration | 76
  Up to D90 : Safety Success | 75
  Up to D180 : No serious dev rel complications | 76
  Up to D180 : No additional surgical intervention | 77
  Up to D180 : No device fracture, migration | 70
  Up to D180 : Safety Success | 70
  Up to D360 : No serious dev rel complications | 74
  Up to D360 : No additional surgical intervention | 74
  Up to D360 : No device fracture, migration | 67
  Up to D360 : Safety Success | 67
Statistical Analysis 1: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 7-14: Subjects who had no serious device related complications; Test type: Other; Percentage of Subjects = 100.0, 95% CI 2-sided [96 to 100]
Statistical Analysis 2: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 7-14: No additional surgical interventions of revisions, supplements, fixations or removals; Test type: Other; Percentage of Subjects = 100, 95% CI 2-sided [96 to 100]
Statistical Analysis 3: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 7-14: Subjects who had no device fracture, migration, mal-alignment or loss of reduction or fixation; Test type: Other; Percentage of Subjects = 98.8, 95% CI 2-sided [93 to 100]
Statistical Analysis 4: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 7-14: Safety Success; Test type: Other; Percentage of Subjects = 98.8, 95% CI 2-sided [93 to 100]
Statistical Analysis 5: Comparison: Photodynamic Bone Stabilization System (PBSS); [analysis description as in outcome 3, analysis 1]; Test type: Other; Percentage of Subjects = 98.8, 95% CI 2-sided [93 to 100]
Statistical Analysis 6: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 30: No additional surgical interventions of revisions, supplements, fixations or removals; Test type: Other; Percentage of Subjects = 98.8, 95% CI 2-sided [93 to 100]
Statistical Analysis 7: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 30: Subjects who had no device fracture, migration, mal-alignment or loss of reduction or fixation; Test type: Other; Percentage of Subjects = 96.3, 95% CI 2-sided [90 to 99]
Statistical Analysis 8: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 30: Safety Success; Test type: Other; Percentage of Subjects = 96.3, 95% CI 2-sided [90 to 99]
Statistical Analysis 9: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 90: Subjects who had no serious device related complications; Test type: Other; Percentage of Subjects = 96.3, 95% CI 2-sided [90 to 99]
Statistical Analysis 10: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 90: No additional surgical interventions of revisions, supplements, fixations or removals; Test type: Other; Percentage of Subjects = 98.8, 95% CI 2-sided [93 to 100]
Statistical Analysis 11: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 90: Subjects who had no device fracture, migration, mal-alignment or loss of reduction or fixation; Test type: Other; Percentage of Subjects = 93.8, 95% CI 2-sided [86 to 98]
Statistical Analysis 12: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 90: Safety Success; Test type: Other; Percentage of Subjects = 92.6, 95% CI 2-sided [85 to 97]
Statistical Analysis 13: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 180: Subjects who had no serious device related complications; Test type: Other; Percentage of Subjects = 93.8, 95% CI 2-sided [86 to 98]
Statistical Analysis 14: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 180: No additional surgical interventions of revisions, supplements, fixations or removals; Test type: Other; Percentage of Subjects = 95.1, 95% CI 2-sided [88 to 99]
Statistical Analysis 15: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 180: Subjects who had no device fracture, migration, mal-alignment or loss of reduction or fixation; Test type: Other; Percentage of Subjects = 86.4, 95% CI 2-sided [77 to 93]
Statistical Analysis 16: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 180: Safety Success; Test type: Other; Percentage of Subjects = 86.4, 95% CI 2-sided [77 to 93]
Statistical Analysis 17: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 360: Subjects who had no serious device related complications; Test type: Other; Percentage of Subjects = 91.4, 95% CI 2-sided [83 to 96]
Statistical Analysis 18: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 360: No additional surgical interventions of revisions, supplements, fixations or removals; Test type: Other; Percentage of Subjects = 91.4, 95% CI 2-sided [83 to 96]
Statistical Analysis 19: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 360: Subjects who had no device fracture, migration, mal-alignment or loss of reduction or fixation; Test type: Other; Percentage of Subjects = 82.7, 95% CI 2-sided [73 to 90]
Statistical Analysis 20: Comparison: Photodynamic Bone Stabilization System (PBSS); 95% exact binomial confidence intervals provided for each of the parameters that make up the safety success endpoint and the safety success endpoint - Up to Day 360: Safety Success; Test type: Other; Percentage of Subjects = 82.7, 95% CI 2-sided [73 to 90]

4. Secondary Outcome: Pain at Palpation
Description: Pain on palpation and clinical significance
Time Frame: 90, 180 and 360 days
Population: Data is presented for subjects who had follow-up visit data. Subjects who withdrew from the study prior to a visit or did not come in for a visit are excluded from the analysis at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Participants
  90 Day F/U: number analyzed (Participants) | 54
  90 Day F/U: Pain on palpation Yes Clinically Si | 4
  90 Day F/U: Pain on palpation Yes Not Clinically Sig | 7
  90 Day F/U: Pain on palpation No | 42
  90 Day F/U: Pain on palpation Not Done | 1
  180 Day F/U: number analyzed (Participants) | 49
  180 Day F/U: Pain on palpation Yes Clinically Si | 8
  180 Day F/U: Pain on palpation Yes Not Clinically Sig | 12
  180 Day F/U: Pain on palpation No | 25
  180 Day F/U: Pain on palpation Not Done | 4
  360 Day F/U: number analyzed (Participants) | 36
  360 Day F/U: Pain on palpation Yes Clinically Si | 3
  360 Day F/U: Pain on palpation Yes Not Clinically Sig | 4
  360 Day F/U: Pain on palpation No | 27
  360 Day F/U: Pain on palpation Not Done | 2

5. Secondary Outcome: Duration of Index Procedure
Description: Duration of index procedure (hours)
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
hours | 1.64 (1.221)

6. Secondary Outcome: Activities of Daily Living Score Through All Follow-up Intervals
Description: Change from Baseline in Activities of Daily Living Score (EORTC QLQ BM22) for each of the four scales at follow-up visits. There are two symptom scales (painful sites and pain characteristics) and two functional scales (functional interface and psychosocial aspects). All scales will be transformed to range in score from 0 to 100. A high score for the symptom scales represented a high level of symptomatology or problems, while a high score for the functional scales represents a high level of functioning.
Time Frame: Baseline, 90, 180 and 360 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
units on a scale
  Functional Interference, 90 Day F/U: number analyzed (Participants) | 55
  Functional Interference, 90 Day F/U | 30.41 (29.362)
  Functional Interference, 180 Day F/U: number analyzed (Participants) | 48
  Functional Interference, 180 Day F/U | 28.86 (33.357)
  Functional Interference, 360 Day F/U: number analyzed (Participants) | 36
  Functional Interference, 360 Day F/U | 35.12 (31.625)
  Psychosocial Aspects, 90 Day F/U: number analyzed (Participants) | 55
  Psychosocial Aspects, 90 Day F/U | 12.73 (22.316)
  Psychosocial Aspects, 180 Day F/U: number analyzed (Participants) | 48
  Psychosocial Aspects, 180 Day F/U | 12.48 (25.522)
  Psychosocial Aspects, 360 Day F/U: number analyzed (Participants) | 36
  Psychosocial Aspects, 360 Day F/U | 16.36 (26.056)
  Painful Sites, 90 Day F/U: number analyzed (Participants) | 55
  Painful Sites, 90 Day F/U | -6.55 (17.093)
  Painful Sites, 180 Day F/U: number analyzed (Participants) | 48
  Painful Sites, 180 Day F/U | -5.56 (17.029)
  Painful Sites, 360 Day F/U: number analyzed (Participants) | 36
  Painful Sites, 360 Day F/U | -5.19 (18.248)
  Pain Characteristics, 90 Day F/U: number analyzed (Participants) | 55
  Pain Characteristics, 90 Day F/U | -32.12 (29.988)
  Pain Characteristics, 180 Day F/U: number analyzed (Participants) | 48
  Pain Characteristics, 180 Day F/U | -28.94 (33.115)
  Pain Characteristics, 360 Day F/U: number analyzed (Participants) | 36
  Pain Characteristics, 360 Day F/U | -37.35 (32.655)

7. Secondary Outcome: MSTS Upper Extremity Functional Outcome
Description: Musculoskeletal Tumor Society Rating Scale for Upper Extremity (MSTS) Functional Outcome. MSTS score is a six-item scale. It ranges from 0 to 30. Higher score is associated with better function. Scores were divided by 30 and multiplied by 100 to facilitate interpretation.
Time Frame: 90, 180, 360 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
units on a scale
  90 Day F/U: number analyzed (Participants) | 52
  90 Day F/U | 40.13 (23.607)
  180 Day F/U: number analyzed (Participants) | 45
  180 Day F/U | 44.15 (26.507)
  360 Day F/U: number analyzed (Participants) | 33
  360 Day F/U | 54.75 (22.608)

8. Secondary Outcome: Assessment of Post-Surgery Status
Description: Number and percent of subjects who receive physical therapy, supportive orthopedic device, or analgesic medication
Time Frame: Surgery & Discharge, 7-14, 30, 90, 180, 360 days
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Participants
  Surgery/Discharge: Physical therapy prescribed | 27
  Surgery/Discharge: Supportive orth dev recommend | 64
  SurgeryDischarge: Analgesic med prescribed | 74
  Surgery/Discharge: Completed physical therapy | NA — Not applicable for this visit
  Surgery/Discharge: Used supportive orth devices | NA — Not applicable for this visit
  Surgery/Discharge: Used analgesic medication | NA — Not applicable for this visit
  7-14 Day F/U: Physical therapy prescribed | 29
  7-14 Day F/U: Supportive orth dev recommend | 28
  7-14 Day F/U: Analgesic medication prescribed | 17
  7-14 Day F/U: Completed physical therapy | 26
  7-14 Day F/U: Used supportive orthopedic devices | 48
  7-14 Day F/U: Used analgesic medication | 64
  30 Day F/U: Physical therapy prescribed | 26
  30 Day F/U: Supportive orth recommend | 13
  30 Day F/U: Analgesic medication prescribed | 19
  30 Day F/U: Completed physical therapy | 32
  30 Day F/U: Used supportive orthopedic devices | 27
  30 Day F/U: Used analgesic medication | 51
  90 Day F/U: Physical therapy prescribed | 17
  90 Day F/U: Supportive orthopedic dev recommend | 6
  90 Day F/U: Analgesic medication prescribed | 8
  90 Day F/U: Completed physical therapy | 31
  90 Day F/U: Used supportive orthopedic devices | 11
  90 Day F/U : Used analgesic medication | 41
  180 Day F/U: Physical therapy prescribed | 12
  180 Day F/U: Supportive orth device recommend | 7
  180 Day F/U: Analgesic medication prescribed | 6
  180 Day F/U: Completed physical therapy | 23
  180 Day F/U: Used supportive orthopedic devices | 4
  180 Day F/U: Used analgesic medication | 33
  360 Day F/U: Physical therapy prescribed | 2
  360 Day F/U: Supportive orth device recommended | 2
  360 Day F/U: Analgesic medication prescribed | 2
  360 Day F/U: Completed physical therapy | 8
  360 Day F/U: Used supportive orthopedic devices | 2
  360 Day F/U: Used analgesic medication | 28

9. Secondary Outcome: Summary of Procedure and Device-Related Complications Rate
Description: Procedure and device-related complications rate presented at follow-up visits
Time Frame: up to day 90, up to day180 since day 90, up to 360 since day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Participants
  Procedure & device-related complications up to D90: During device preparation | 0
  Procedure & device-related complications up to D90: During device implantation | 1
  Procedure & device-related complications up to D90: Post-implantation | 3
  Procedure & device-related complications up to D90: None | 77
  Proc & dev-related comp rate up D180 since D90: During device preparation | NA — Post-op visit
  Proc & dev-related comp rate up D180 since D90: During device implantation | NA — Post-op visit
  Proc & dev-related comp rate up D180 since D90: Post-implantation | 6
  Proc & dev-related comp rate up D180 since D90: None | 75
  Proc & dev-related comp rate up to D360 since D180: During device preparation | NA — Post-op visit
  Proc & dev-related comp rate up to D360 since D180: During device implantation | NA — Post-op visit
  Proc & dev-related comp rate up to D360 since D180: Post-implantation | 4
  Proc & dev-related comp rate up to D360 since D180: None | 77

10. Secondary Outcome: Summary of Change From Baseline Range of Motion by Visit and Test
Description: Range of motions tests (abduction, extension, flexion, lateral rotation and medial rotation) for active range of motion and passive range of motion for the affected and unaffected arm.
Time Frame: Baseline, 90, 180 and 360 Days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
degrees
  90 Day F/U, Abduction, Active ROM affected arm: number analyzed (Participants) | 44
  90 Day F/U, Abduction, Active ROM affected arm | 31.3 (33.36)
  90 Day F/U, Abduction, Passive ROM affected arm: number analyzed (Participants) | 42
  90 Day F/U, Abduction, Passive ROM affected arm | 29.1 (38.22)
  180 Day F/U, Abduction, Active ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U, Abduction, Active ROM affected arm | 41.0 (36.04)
  180 Day F/U Abduction, Passive ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U Abduction, Passive ROM affected arm | 31.2 (37.71)
  360 Day F/U, Abduction, Active ROM affected arm: number analyzed (Participants) | 31
  360 Day F/U, Abduction, Active ROM affected arm | 54.9 (44.42)
  360 Day F/U, Abduction, Passive ROM affected arm: number analyzed (Participants) | 32
  360 Day F/U, Abduction, Passive ROM affected arm | 46.3 (51.24)
  90 Day F/U, Abduction, Active ROM unaffected arm: number analyzed (Participants) | 32
  90 Day F/U, Abduction, Active ROM unaffected arm | 2 (32.14)
  90 Day F/U, Abduction, Pass ROM unaffected arm: number analyzed (Participants) | 30
  90 Day F/U, Abduction, Pass ROM unaffected arm | -0.5 (29.19)
  180 Day F/U, Abduction, Active ROM unaffected arm: number analyzed (Participants) | 26
  180 Day F/U, Abduction, Active ROM unaffected arm | 4.9 (33.29)
  180 Day F/U, Abduction, Passive ROM unaffected arm: number analyzed (Participants) | 26
  180 Day F/U, Abduction, Passive ROM unaffected arm | 6.0 (32.46)
  360 Day F/U, Abduction, Active ROM unaffected arm: number analyzed (Participants) | 25
  360 Day F/U, Abduction, Active ROM unaffected arm | 19.1 (43.62)
  360 Day F/U, Abduction, Passive ROM unaffected arm: number analyzed (Participants) | 24
  360 Day F/U, Abduction, Passive ROM unaffected arm | 16.0 (42.13)
  90 Day F/U, Extension, Active ROM affected arm: number analyzed (Participants) | 43
  90 Day F/U, Extension, Active ROM affected arm | 12 (14.88)
  90 Day F/U, Extension, Passive ROM affected arm: number analyzed (Participants) | 40
  90 Day F/U, Extension, Passive ROM affected arm | 11.7 (17.01)
  180 Day F/U, Extension, Active ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U, Extension, Active ROM affected arm | 8.1 (16.17)
  180 Day F/U, Extension, Passive ROM affected arm: number analyzed (Participants) | 36
  180 Day F/U, Extension, Passive ROM affected arm | 4.8 (17.15)
  360 Day F/U, Extension, Active ROM affected arm: number analyzed (Participants) | 31
  360 Day F/U, Extension, Active ROM affected arm | 10.3 (19.75)
  360 Day F/U, Extension, Passive ROM affected arm: number analyzed (Participants) | 31
  360 Day F/U, Extension, Passive ROM affected arm | 7.7 (21.83)
  90 Day F/U, Extension, Active ROM unaffected arm: number analyzed (Participants) | 31
  90 Day F/U, Extension, Active ROM unaffected arm | 0.6 (13.87)
  90 Day F/U, Extension, Passive ROM unaffected arm: number analyzed (Participants) | 29
  90 Day F/U, Extension, Passive ROM unaffected arm | -1.0 (14.12)
  180 Day F/U, Extension, Active ROM unaffected arm: number analyzed (Participants) | 25
  180 Day F/U, Extension, Active ROM unaffected arm | -4.1 (17.96)
  180 Day F/U, Extension, Passive ROM unaffected arm: number analyzed (Participants) | 25
  180 Day F/U, Extension, Passive ROM unaffected arm | -4.1 (17.41)
  360 Day F/U, Extension, Active ROM unaffected arm: number analyzed (Participants) | 24
  360 Day F/U, Extension, Active ROM unaffected arm | 3.5 (19.90)
  360 Day F/U, Extension, Passive ROM unaffected arm: number analyzed (Participants) | 23
  360 Day F/U, Extension, Passive ROM unaffected arm | 5.5 (27.24)
  90 Day F/U, Flexion, Active ROM affected arm: number analyzed (Participants) | 43
  90 Day F/U, Flexion, Active ROM affected arm | 28.7 (36.61)
  90 Day F/U, Flexion, Passive ROM affected arm: number analyzed (Participants) | 42
  90 Day F/U, Flexion, Passive ROM affected arm | 28.5 (45.27)
  180 Day F/U, Flexion, Active ROM affected arm: number analyzed (Participants) | 36
  180 Day F/U, Flexion, Active ROM affected arm | 33.1 (39.90)
  180 Day F/U, Flexion, Passive ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U, Flexion, Passive ROM affected arm | 29.4 (45.35)
  360 Day F/U, Flexion, Active ROM affected arm: number analyzed (Participants) | 30
  360 Day F/U, Flexion, Active ROM affected arm | 46.6 (51.17)
  360 Day F/U, Flexion, Passive ROM affected arm: number analyzed (Participants) | 32
  360 Day F/U, Flexion, Passive ROM affected arm | 36.7 (52.28)
  90 Day F/U, Flexion, Active ROM unaffected arm: number analyzed (Participants) | 32
  90 Day F/U, Flexion, Active ROM unaffected arm | 5.6 (29.85)
  90 Day F/U, Flexion, Passive ROM unaffected arm: number analyzed (Participants) | 30
  90 Day F/U, Flexion, Passive ROM unaffected arm | 3.7 (29.02)
  180 Day F/U, Flexion, Active ROM unaffected arm: number analyzed (Participants) | 26
  180 Day F/U, Flexion, Active ROM unaffected arm | 3.0 (35.86)
  180 Day F/U, Flexion, Passive ROM unaffected arm: number analyzed (Participants) | 26
  180 Day F/U, Flexion, Passive ROM unaffected arm | 1.8 (34.72)
  360 Day F/U, Flexion, Active ROM unaffected arm: number analyzed (Participants) | 25
  360 Day F/U, Flexion, Active ROM unaffected arm | 7.5 (42.01)
  360 Day F/U, Flexion, Passive ROM unaffected arm: number analyzed (Participants) | 24
  360 Day F/U, Flexion, Passive ROM unaffected arm | 4.7 (41.50)
  90 Day F/U, Lat Rotate, Active ROM affected arm: number analyzed (Participants) | 44
  90 Day F/U, Lat Rotate, Active ROM affected arm | 10.4 (22.51)
  90 Day F/U, Lat Rotate, Passive ROM affected arm: number analyzed (Participants) | 42
  90 Day F/U, Lat Rotate, Passive ROM affected arm | 8.6 (23.61)
  180 Day F/U, Lat Rotate, Active ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U, Lat Rotate, Active ROM affected arm | 12.4 (31.38)
  180 Day F/U, Lat Rotate, Passive ROM affected arm: number analyzed (Participants) | 37
  180 Day F/U, Lat Rotate, Passive ROM affected arm | 6.5 (30.69)
  360 Day F/U, Lat Rotate, Active ROM affected arm: number analyzed (Participants) | 31
  360 Day F/U, Lat Rotate, Active ROM affected arm | 16.6 (22.79)
  360 Day F/U, Lat Rotate, Passive ROM affected arm: number analyzed (Participants) | 32
  360 Day F/U, Lat Rotate, Passive ROM affected arm | 13.6 (20.99)
  90 Day F/U, Lat Rotate, Active ROM unaffected arm: number analyzed (Participants) | 31
  90 Day F/U, Lat Rotate, Active ROM unaffected arm | 0.5 (14.95)
  90 Day F/U, Lat Rotate, Passive ROM unaffected arm: number analyzed (Participants) | 29
  90 Day F/U, Lat Rotate, Passive ROM unaffected arm | 0.3 (14.18)
  180 Day F/U, Lat Rotate, Active ROM unaffected arm: number analyzed (Participants) | 25
  180 Day F/U, Lat Rotate, Active ROM unaffected arm | -3.6 (18.67)
  180 Day F/U, Lat Rotate, Passive ROM unaffect arm: number analyzed (Participants) | 25
  180 Day F/U, Lat Rotate, Passive ROM unaffect arm | -6.0 (19.14)
  360 Day F/U, Lat Rotate, Active ROM unaffected arm: number analyzed (Participants) | 24
  360 Day F/U, Lat Rotate, Active ROM unaffected arm | 1.8 (20.25)
  360 Day F/U, Lat Rotate, Passive ROM unaffect arm: number analyzed (Participants) | 23
  360 Day F/U, Lat Rotate, Passive ROM unaffect arm | -0.22 (25.656)
  90 Day F/U, Med Rotate, Active ROM affected arm: number analyzed (Participants) | 41
  90 Day F/U, Med Rotate, Active ROM affected arm | 11.7 (28.78)
  90 Day F/U, Med Rotate, Passive ROM affected arm: number analyzed (Participants) | 39
  90 Day F/U, Med Rotate, Passive ROM affected arm | 7.5 (25.90)
  180 Day F/U, Med Rotate, Active ROM affected arm: number analyzed (Participants) | 36
  180 Day F/U, Med Rotate, Active ROM affected arm | 2.2 (31.21)
  180 Day F/U, Med Rotate, Passive ROM affected arm: number analyzed (Participants) | 36
  180 Day F/U, Med Rotate, Passive ROM affected arm | 3.1 (34.14)
  360 Day F/U, Med Rotate, Active ROM affected arm: number analyzed (Participants) | 31
  360 Day F/U, Med Rotate, Active ROM affected arm | 6.4 (27.46)
  360 Day F/U, Med Rotate, Passive ROM affected arm: number analyzed (Participants) | 32
  360 Day F/U, Med Rotate, Passive ROM affected arm | 6.3 (24.28)
  90 Day F/U, Med Rotate, Active ROM unaffected arm: number analyzed (Participants) | 30
  90 Day F/U, Med Rotate, Active ROM unaffected arm | 1.7 (14.43)
  90 Day F/U, Med Rotate, Passive ROM unaffected arm: number analyzed (Participants) | 28
  90 Day F/U, Med Rotate, Passive ROM unaffected arm | 2.89 (20.939)
  180 Day F/U, Med Rotate, Active ROM unaffected arm: number analyzed (Participants) | 24
  180 Day F/U, Med Rotate, Active ROM unaffected arm | -1.3 (14.72)
  180 Day F/U, Med Rotate, Passive ROM unaffect arm: number analyzed (Participants) | 24
  180 Day F/U, Med Rotate, Passive ROM unaffect arm | 0.8 (9.85)
  360 Day F/U, Med Rotate, Active ROM unaffected arm: number analyzed (Participants) | 23
  360 Day F/U, Med Rotate, Active ROM unaffected arm | 2.6 (19.15)
  360 Day F/U, Med Rotate, Passive ROM unaffect arm: number analyzed (Participants) | 22
  360 Day F/U, Med Rotate, Passive ROM unaffect arm | 2.5 (18.76)

11. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay (from day of procedure to day of discharge)
Time Frame: From day of procedure until the day of hospital discharge (up to 36 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
Number analyzed (Participants) | 81
Days | 5.1 (6.14)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Photodynamic Bone Stabilization System (PBSS)
All-Cause Mortality (participants affected / at risk) | 32/81
Serious Adverse Events (participants affected / at risk) | 58/81
Other Adverse Events (participants affected / at risk) | 49/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Bone Stabilization System (PBSS) (N=81)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Medical device site pain (General disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chondrosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endotheliomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device breakage (Product Issues) | 7 (7)
Device dislocation (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photodynamic Bone Stabilization System (PBSS) (N=81)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Medical device site pain (General disorders) | 3 (3)
Medical device site swelling (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Haemoglobin decreased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone lesion (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Device breakage (Product Issues) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall submit copies of any material to sponsor for review at least 30 days in advance of submission to a publisher or other third party. The sponsor shall review the data provided for consistency and reserves the right to delete any confidential information or other proprietary information from the proposed material. Sponsor may extend such review period for another 60 days to allow for filing of patent applications or take other steps to protect the sponsor's IP interests.

DOCUMENTS (2):
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT02338492/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02338492/SAP_001.pdf